CLINICAL TRIAL: NCT00002537
Title: A PHASE I STUDY OF PROLONGED LOW-DOSE TOPOTECAN INFUSION COMBINED WITH CHEST IRRADIATION
Brief Title: Radiation Therapy Plus Topotecan in Treating Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02487; NYU-9301; NCI-T93-0015D; CDR0000078480 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2006-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Topotecan; Radiotherapy

ARMS (1):
- Arm I (Experimental): Beginning on day 1, patients receive topotecan IV continuously for 3-6 weeks and thoracic radiotherapy 5 days a week for 2, 3, or 6 weeks. Cohorts of 4-6 patients receive escalating doses of topotecan and thoracic radiotherapy until the maximum tolerated dose (MTD) of each therapy is determined. The MTD is defined as the dose preceding that at which 2 of 4 or 6 patients experience dose-limiting toxicity. Six additional patients are treated at the MTD. Patients who fail to achieve complete remission (CR) and continue to have measurable disease at 4-6 weeks after completion of radiotherapy receive topotecan IV continuously on days 1-21 at 1 dose level preceding the MTD as determined by the ongoing Protocol NYU-9123. Treatment continues every 4 weeks in the absence of unacceptable toxicity.
  Interventions: Drug: topotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Drug: topotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
Phase I trial to study the effectiveness of radiation therapy plus topotecan in treating patients who have non-small cell lung cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of topotecan and chest irradiation in patients with non-small cell lung cancer.

II. Determine the qualitative and quantitative toxic effects of this regimen in these patients.

III. Determine the degree of antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation study of topotecan and thoracic radiotherapy.

Beginning on day 1, patients receive topotecan IV continuously for 3-6 weeks and thoracic radiotherapy 5 days a week for 2, 3, or 6 weeks. Cohorts of 4-6 patients receive escalating doses of topotecan and thoracic radiotherapy until the maximum tolerated dose (MTD) of each therapy is determined. The MTD is defined as the dose preceding that at which 2 of 4 or 6 patients experience dose-limiting toxicity. Six additional patients are treated at the MTD. Patients who fail to achieve complete remission (CR) and continue to have measurable disease at 4-6 weeks after completion of radiotherapy receive topotecan IV continuously on days 1-21 at 1 dose level preceding the MTD as determined by the ongoing Protocol NYU-9123. Treatment continues every 4 weeks in the absence of unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven non-small cell lung cancer
* Eligible for chest irradiation with 3,000 to 6,000 cGy (based upon standard radiotherapy indications)
* Measurable or evaluable disease
* Measurable disease defined as bidimensionally measurable lesion on physical exam or radiograph (CT or MRI acceptable)

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: 0-2
* Life expectancy: At least 12 weeks
* WBC at least 4,000/mm3
* Platelet count at least 100,000/mm3
* Bilirubin no greater than 1.5 mg/dL
* AST less than 3 times normal
* Alkaline phosphatase less than 3 times normal
* Creatinine no greater than 1.5 mg/dL
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* No more than 1 prior chemotherapy regimen allowed
* At least 4 weeks since prior chemotherapy and recovered
* No prior radiotherapy
* Recovered from toxic effects of any prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1993-09; Primary Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States